CLINICAL TRIAL: NCT00433030
Title: Observational Cohort of HIV Infected Adults and Children in the PHPT Network Hospitals in Thailand
Status: Completed | Type: Observational
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Global Fund (Other); Ministry of Health, Thailand (Other Government)
Responsible Party: Principal Investigator, GONZAGUE JOURDAIN, Senior Researcher, Institut de Recherche pour le Developpement
Other Study IDs: PHPT-Cohort
Record Dates: First submitted 2007-02-08; First posted 2007-02-09 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: HIV Infections
Keywords: Highly Active Antiretroviral Therapy; HIV Viral load; HIV drug Resistance; Thailand
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Since 2004, the Thai Ministry of Public Health has massively scaled up antiretroviral treatment programs to provide therapy to more than 80,000 patients with partial support of the Global Fund to fight AIDS, Tuberculosis and Malaria (GFATM).

As access to HIV care continues to expand under the universal health coverage system, it is important to document and analyze the efficacy, tolerance, toxicity and acceptability of antiretroviral therapy within pilot treatment programs, to provide evidence based feedback and recommendations to the national program and policy makers.

DETAILED DESCRIPTION:
As Thailand is rapidly expanding access to antiretroviral treatments under the universal health coverage system, it is crucial to document and learn from pilot antiretroviral treatment programs, in particular the medical outcomes and logistical, and organizational issues faced by hospital teams and patients in order to adapt the ARV delivery and monitoring system to various local settings.

Specific objectives

1. Analyze data collected in patients participating in the PHPT antiretroviral treatment program, in accordance to national and international guidelines, with no experimental interventions.
2. To determine factors associated with treatment outcome including immune status, virologic factors and antiretroviral drugs levels
3. To study the operational aspects of integrating comprehensive HIV care into the existing care system with regards to new activities generated at the hospital level (counseling, referral systems, biological monitoring), the impact on other health activities, mobilization of human and financial resources, affordability and sustainability.

The population of the study consists of approximately 2,000 consenting HIV-infected patients, including one-third of children, receiving HIV care as part of the GF-ATM or OXFAM Access to Antiretroviral programs, presenting at any of the PHPT network hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Adults and children (children are defined as less than 18 years old) patients are eligible for the inclusion in the cohort if they meet all the following inclusion criteria:

  * Participation in the GFATM or Oxfam Access to Antiretroviral Programs
  * For adults, consent to have their clinical or biological data used for this research study, and willingness to be followed at one of the PHPT network hospitals. For children, caregiver's consent to participate, willingness to bring the child to the scheduled visits for the duration of the treatment, and to have the child's clinical or biological data used for this research study.

Exclusion Criteria:

* This is an observational study of an access to treatment program, therefore all patients who require treatment and are willing to be followed by the medical team and have their data collected can be enrolled in the study. The only exclusion criteria would be refusal to participate and the discontinuation criteria would be withdrawal of consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-infected Adults and Children
Sampling Method: Non-Probability Sample
Enrollment: 2816 (Actual)
Dates: Start 2007-01; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gonzague JOURDAIN, MD, PhD, Principal Investigator — Institut de Recherche pour le Developpement
Locations (38):
- Thailand (38):
  - Mae Chan Hospital, Mae Chan, Changwat Chiang Rai
  - Mae Sai Hospital, Mae Sai, Changwat Chiang Rai
  - Phan Hospital, Phan, Changwat Chiang Rai
  - Somdej Pranangchao Sirikit Hospital, Sattahip, Changwat Chon Buri
  - Kranuan Crown Prince Hospital, Kranuan, Changwat Khon Kaen
  - Chiang Kham Hospital, Chiang Kham, Changwat Phayao
  - Hat Yai Hospital, Hat Yai, Changwat Songkhla
  - Doi Saket Hospital, Doi Saket, Chiang Mai
  - Mae on Hospital, Mae On, Chiang Mai
  - Nakornping Hospital, Mae Rim, Chiang Mai
  - San Kamphaeng Hospital, San Kamphaeng, Chiang Mai
  - Sanpatong Hospital, San Pa Tong, Chiang Mai
  - San Sai Hospital, San Sai, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai, Chiangrai
  - Mahasarakam Hospital, Maha Sarakham, Mahasarakam
  - Nakhonpathom Hospital, Nakhon Pathom, Nakhonpathom
  - Bhumibol Adulyadej Hospital, Bangkok
  - Nopparat Rajathanee Hospital, Bangkok
  - Somdej Prapinklao Hospital, Bangkok
  - Chacheongsao Hospital, Chachoengsao
  - Prapokklao Hospital, Chanthaburi
  - Chonburi Hospital, Chon Buri
  - Kalasin Hospital, Kalasin
  - Phaholpolphayuhasena Hospital, Kanchanaburi
  - Khon Kaen Hospital, Khon Kaen
  - Regional Health Promotion Centre 6, Khon Kaen, Khon Kaen
  - Lampang Hospital, Lampang
  - Lamphun Hospital, Lamphun
  - Samutprakarn Hospital, Mueang Samut Prakan
  - Maharaj Nakornratchasrima Hospital, Nakhon Ratchasima
  - Nong Khai Hospital, Nong Khai
  - Pranangklao Hospital, Nonthaburi
  - Phayao Provincial Hospital, Phayao
  - Buddhachinaraj Hospital, Phitsanulok
  - Ratchaburi Hospital, Ratchaburi
  - Rayong Hospital, Rayong
  - Roi-et Hospital, Roi Et
  - Samutsakon Hospital, Samut Sakhon

REFERENCES:
- [Result] Collins IJ, Jourdain G, Hansudewechakul R, Kanjanavanit S, Hongsiriwon S, Ngampiyasakul C, Sriminiphant S, Technakunakorn P, Ngo-Giang-Huong N, Duong T, Le Coeur S, Jaffar S, Lallemant M; Program for HIV Prevention and Treatment Study Team. Long-term survival of HIV-infected children receiving antiretroviral therapy in Thailand: a 5-year observational cohort study. Clin Infect Dis. 2010 Dec 15;51(12):1449-57. doi: 10.1086/657401. Epub 2010 Nov 5. PMID 21054181
- [Result] Ngo-Giang-Huong N, Jourdain G, Amzal B, Sang-a-gad P, Lertkoonalak R, Eiamsirikit N, Tansuphasawasdikul S, Buranawanitchakorn Y, Yutthakasemsunt N, Mekviwattanawong S, McIntosh K, Lallemant M; Program for HIV Prevention and Treatment (PHPT) study group. Resistance patterns selected by nevirapine vs. efavirenz in HIV-infected patients failing first-line antiretroviral treatment: a bayesian analysis. PLoS One. 2011;6(11):e27427. doi: 10.1371/journal.pone.0027427. Epub 2011 Nov 23. PMID 22132100
- [Result] Jourdain G, Wagner TA, Ngo-Giang-Huong N, Sirirungsi W, Klinbuayaem V, Fregonese F, Nantasen I, Techapornroong M, Halue G, Nilmanat A, Wittayapraparat P, Chalermpolprapa V, Pathipvanich P, Yuthavisuthi P, Frenkel LM, Lallemant M; Program for HIV Prevention and Treatment (PHPT) Study Group. Association between detection of HIV-1 DNA resistance mutations by a sensitive assay at initiation of antiretroviral therapy and virologic failure. Clin Infect Dis. 2010 May 15;50(10):1397-404. doi: 10.1086/652148. PMID 20377404
- [Result] Wagner TA, Kress CM, Beck I, Techapornroong M, Wittayapraparat P, Tansuphasawasdikul S, Jourdain G, Ngo-Giang-Huong N, Lallemant M, Frenkel LM. Detection of HIV-1 drug resistance in women following administration of a single dose of nevirapine: comparison of plasma RNA to cellular DNA by consensus sequencing and by oligonucleotide ligation assay. J Clin Microbiol. 2010 May;48(5):1555-61. doi: 10.1128/JCM.02062-09. Epub 2010 Feb 24. PMID 20181911
- [Result] Fregonese F, Collins IJ, Jourdain G, Lecoeur S, Cressey TR, Ngo-Giang-Houng N, Banchongkit S, Chutanunta A, Techapornroong M, Lallemant M; Program for HIV Prevention and Treatment Study Group. Predictors of 5-year mortality in HIV-infected adults starting highly active antiretroviral therapy in Thailand. J Acquir Immune Defic Syndr. 2012 May 1;60(1):91-8. doi: 10.1097/QAI.0b013e31824bd33f. PMID 22293548
- [Result] Duong T, Jourdain G, Ngo-Giang-Huong N, Le Coeur S, Kantipong P, Buranabanjasatean S, Leenasirimakul P, Ariyadej S, Tansuphasawasdikul S, Thongpaen S, Lallemant M; Program for HIV Prevention and Treatment Study Group. Laboratory and clinical predictors of disease progression following initiation of combination therapy in HIV-infected adults in Thailand. PLoS One. 2012;7(8):e43375. doi: 10.1371/journal.pone.0043375. Epub 2012 Aug 15. PMID 22905264
- [Result] Khamduang W, Gaudy-Graffin C, Ngo-Giang-Huong N, Jourdain G, Moreau A, Luekamlung N, Halue G, Buranawanitchakorn Y, Kunkongkapan S, Buranabanjasatean S, Lallemant M, Sirirungsi W, Goudeau A; Program for HIV Prevention and Treatment Study Group. Long-term hepatitis B virus (HBV) response to lamivudine-containing highly active antiretroviral therapy in HIV-HBV co-infected patients in Thailand. PLoS One. 2012;7(7):e42184. doi: 10.1371/journal.pone.0042184. Epub 2012 Jul 31. PMID 22860080
- [Result] Collins IJ, Cairns J, Jourdain G, Fregonese F, Nantarukchaikul M, Lertpienthum N, Wannarit P, Attavinijtrakarn P, Layangool P, Le Coeur S, Lallemant M; Program for HIV Prevention and Treatment (PHPT) study team. Hospitalization trends, costs, and risk factors in HIV-infected children on antiretroviral therapy. AIDS. 2012 Sep 24;26(15):1943-52. doi: 10.1097/QAD.0b013e328357f7b9. PMID 22824633
- [Result] Puthanakit T, Jourdain G, Hongsiriwon S, Suntarattiwong P, Chokephaibulkit K, Sirisanthana V, Kosalaraksa P, Petdachai W, Hansudewechakul R, Siangphoe U, Suwanlerk T, Ananworanich J; HIV-NAT 086Study Team. HIV-1 drug resistance mutations in children after failure of first-line nonnucleoside reverse transcriptase inhibitor-based antiretroviral therapy. HIV Med. 2010 Oct 1;11(9):565-72. doi: 10.1111/j.1468-1293.2010.00828.x. Epub 2010 Mar 25. PMID 20345882
- [Result] Sukasem C, Cressey TR, Prapaithong P, Tawon Y, Pasomsub E, Srichunrusami C, Jantararoungtong T, Lallement M, Chantratita W. Pharmacogenetic markers of CYP2B6 associated with efavirenz plasma concentrations in HIV-1 infected Thai adults. Br J Clin Pharmacol. 2012 Dec;74(6):1005-12. doi: 10.1111/j.1365-2125.2012.04288.x. PMID 22471906
- [Result] Puthanakit T, Jourdain G, Suntarattiwong P, Chokephaibulkit K, Siangphoe U, Suwanlerk T, Prasitsuebsai W, Sirisanthana V, Kosalaraksa P, Petdachai W, Hansudewechakul R, Waranawat N, Ananworanich J; HIV-NAT 086 study team. High virologic response rate after second-line boosted protease inhibitor-based antiretroviral therapy regimens in children from a resource limited setting. AIDS Res Ther. 2012 Jun 18;9(1):20. doi: 10.1186/1742-6405-9-20. PMID 22709957
- [Result] Collins I, Cairns J, Le Coeur S, Pagdi K, Ngampiyaskul C, Layangool P, Borkird T, Na-Rajsima S, Wanchaitanawong V, Jourdain G, Lallemant M. Five-year trends in antiretroviral usage and drug costs in HIV-infected children in Thailand. J Acquir Immune Defic Syndr. 2013 Sep 1;64(1):95-102. doi: 10.1097/QAI.0b013e318298a309. PMID 23945253
- [Result] Tang MW, Rhee SY, Bertagnolio S, Ford N, Holmes S, Sigaloff KC, Hamers RL, de Wit TF, Fleury HJ, Kanki PJ, Ruxrungtham K, Hawkins CA, Wallis CL, Stevens W, van Zyl GU, Manosuthi W, Hosseinipour MC, Ngo-Giang-Huong N, Belec L, Peeters M, Aghokeng A, Bunupuradah T, Burda S, Cane P, Cappelli G, Charpentier C, Dagnra AY, Deshpande AK, El-Katib Z, Eshleman SH, Fokam J, Gody JC, Katzenstein D, Koyalta DD, Kumwenda JJ, Lallemant M, Lynen L, Marconi VC, Margot NA, Moussa S, Ndung'u T, Nyambi PN, Orrell C, Schapiro JM, Schuurman R, Sirivichayakul S, Smith D, Zolfo M, Jordan MR, Shafer RW. Nucleoside reverse transcriptase inhibitor resistance mutations associated with first-line stavudine-containing antiretroviral therapy: programmatic implications for countries phasing out stavudine. J Infect Dis. 2013 Jun 15;207 Suppl 2(Suppl 2):S70-7. doi: 10.1093/infdis/jit114. PMID 23687292
- [Result] Collins IJ, Cairns J, Ngo-Giang-Huong N, Sirirungsi W, Leechanachai P, Le Coeur S, Samleerat T, Kamonpakorn N, Mekmullica J, Jourdain G, Lallemant M; Programme for HIV Prevention and Treatment Study Team. Cost-effectiveness of early infant HIV diagnosis of HIV-exposed infants and immediate antiretroviral therapy in HIV-infected children under 24 months in Thailand. PLoS One. 2014 Mar 14;9(3):e91004. doi: 10.1371/journal.pone.0091004. eCollection 2014. PMID 24632750
- [Result] Suaysod R, Ngo-Giang-Huong N, Salvadori N, Cressey TR, Kanjanavanit S, Techakunakorn P, Krikajornkitti S, Srirojana S, Laomanit L, Chalermpantmetagul S, Lallemant M, Le Coeur S, McIntosh K, Traisathit P, Jourdain G. Treatment Failure in HIV-Infected Children on Second-line Protease Inhibitor-Based Antiretroviral Therapy. Clin Infect Dis. 2015 Jul 1;61(1):95-101. doi: 10.1093/cid/civ271. Epub 2015 Apr 1. PMID 25838288
- [Result] Riyaten P, Salvadori N, Traisathit P, Ngo-Giang-Huong N, Cressey TR, Leenasirimakul P, Techapornroong M, Bowonwatanuwong C, Kantipong P, Nilmanat A, Yutthakasemsunt N, Chutanunta A, Thongpaen S, Klinbuayaem V, Decker L, Le Coeur S, Lallemant M, Capeau J, Mary JY, Jourdain G. New-Onset Diabetes and Antiretroviral Treatments in HIV-Infected Adults in Thailand. J Acquir Immune Defic Syndr. 2015 Aug 1;69(4):453-9. doi: 10.1097/QAI.0000000000000647. PMID 25886928
- [Result] Traisathit P, Delory T, Ngo-Giang-Huong N, Somsamai R, Techakunakorn P, Theansavettrakul S, Kanjanavanit S, Mekmullica J, Ngampiyaskul C, Na-Rajsima S, Lallemant M, Cressey TR, Jourdain G, Collins IJ, Le Coeur S. Brief Report: AIDS-Defining Events and Deaths in HIV-Infected Children and Adolescents on Antiretrovirals: A 14-Year Study in Thailand. J Acquir Immune Defic Syndr. 2018 Jan 1;77(1):17-22. doi: 10.1097/QAI.0000000000001571. PMID 29040162
- [Result] Delory T, Ngo-Giang-Huong N, Rangdaeng S, Chotivanich N, Limtrakul A, Putiyanun C, Suriyachai P, Matanasarawut W, Jarupanich T, Liampongsabuddhi P, Heard I, Jourdain G, Lallemant M, Le Coeur S; PapilloV study group. Human Papillomavirus infection and cervical lesions in HIV infected women on antiretroviral treatment in Thailand. J Infect. 2017 May;74(5):501-511. doi: 10.1016/j.jinf.2017.02.007. Epub 2017 Feb 28. PMID 28254419
- [Result] Salvadori N, Ngo-Giang-Huong N, Duclercq C, Kanjanavanit S, Ngampiyaskul C, Techakunakorn P, Puangsombat A, Figoni J, Mary JY, Collins IJ, Cressey TR, Le Coeur S, Sirirungsi W, Lallemant M, McIntosh K, Jourdain G. Incidence of Tuberculosis and Associated Mortality in a Cohort of Human Immunodeficiency Virus-Infected Children Initiating Antiretroviral Therapy. J Pediatric Infect Dis Soc. 2017 Jun 1;6(2):161-167. doi: 10.1093/jpids/piw090. PMID 28204517
- [Result] Homkham N, Cressey TR, Ingsrisawang L, Bouazza N, Ngampiyaskul C, Hongsiriwon S, Srirojana S, Kanjanavanit S, Bhakeecheep S, Coeur SL, Salvadori N, Treluyer JM, Jourdain G, Urien S. A Population Pharmacokinetic/Pharmacodynamic Model Predicts Favorable HDL Cholesterol Changes Over the First 5 Years in Children Treated With Current Efavirenz-Based Regimens. J Clin Pharmacol. 2016 Sep;56(9):1076-83. doi: 10.1002/jcph.701. Epub 2016 Feb 24. PMID 26749102
- [Result] European Pregnancy and Paediatric HIV Cohort Collaboration (EPPICC) Study Group in EuroCoord. Safety of darunavir and atazanavir in HIV-infected children in Europe and Thailand. Antivir Ther. 2016;21(4):353-8. doi: 10.3851/IMP3008. Epub 2015 Nov 12. PMID 26561496
- [Derived] Kawilapat S, Salvadori N, Ngo-Giang-Huong N, Decker L, Kanjanavanit S, Puangsombat A, Preedisripipat K, Lertpienthum N, Akarathum N, Mekmullica J, Srirompotong U, Lallemant M, Le Coeur S, Traisathit P, Leroi C, Jourdain G. Incidence and risk factors of loss to follow-up among HIV-infected children in an antiretroviral treatment program. PLoS One. 2019 Sep 17;14(9):e0222082. doi: 10.1371/journal.pone.0222082. eCollection 2019. PMID 31527875